CLINICAL TRIAL: NCT02663180
Title: Effects of an Educational Program on Depression Literacy and Stigma Among Students of Secondary Schools in Jazan City
Brief Title: Effects of an Educational Program on Depression Literacy and Stigma Among Secondary School Students in Jazan City
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jazan (Other Government)
Collaborators: Saudi Board of Community Medicine (Unknown)
Responsible Party: Principal Investigator, Hussain Darraj, Community Medicine physician, Ministry of Health, Saudi Arabia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: U1111-1179-1857
Record Dates: First submitted 2016-01-19; First posted 2016-01-26 (Estimated); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Depression Literacy; Depression Stigma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): they will be enrolled in an educational program and video contact.
  Interventions: Behavioral: Educational program; Behavioral: Video contact
- Control group (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Educational program — Educational strategies: 2 Lecture about depression 30 minutes supported by group discussion, brochures and display of posters with mental-health slogans on depression in the schools.
  Arms: Intervention group
Behavioral: Video contact — Contact strategies: Investigators will show a video of a young male who had been diagnosed with depression. The video presented information that was moderately disconfirming of prior stereotypes by balancing the individual's difficulties resulting from Depression, with his ability to live a normal life.
  Arms: Intervention group

SUMMARY:
Depression is a serious mental health disease. It is generally characterized by sadness, loss of interest in activities, and decreased energy. Globally, it is estimated that almost 350 million people suffer from depression. In Saudi Arabia, literature suggested that prevalence of depression among boy's secondary school students in Abha city was 38.2%. Another study found that the prevalence of depression was 22.4 % as moderate, 7.3 % as severe and 3.7% as very severe, with a clear predominance prevalence of depression in girls as in boys (1.5 times). It is important to assess depression literacy including knowledge and beliefs about mental disorders among adolescent. A high level of mental health literacy on depression leads to a better understanding and outcomes of depressive disorders. Schools are a typical venue in which to embed mental health literacy because the school students are more familiar with educational activities. Studies concluded that educational intervention about depression literacy and destigmatization improves knowledge and may decrease stigma. Further research, intervention and activism are needed in the field of mental health in Arab countries to improve awareness of mental health problems.

Objectives: This study is aimed to measure the effect of educational intervention program about depression among secondary schools in Jazan city on depression literacy and stigma during the academic year 2015-2016.

The intervention: the intervention will held at each selected intervention school separately. The program will be over 2 weeks intervention as the following:

* Educational strategies: 2 Lecture about depression 30 minutes supported by group discussion, brochures and display of posters with mental-health slogans on depression in the schools.
* Contact strategies: the investigators will show a video of a young male who had been diagnosed (i.e., not an actor) with depression.

Benefits:

* The intervention group will join educational intervention program they expected to benefit from the program through increase their depression literacy and improve depression stigma, and control group will not join any form of intervention.

Risk: There is no expected risk for participating in the study.

Consent: Three Informed Consents forms will be signed from students, guardians and school manager.

ELIGIBILITY:
Inclusion Criteria:

* Students needed to be enrolled in one of the selected schools during the academic year 2015-2016.
* Must be in the age group 10-19 years.
* Must agree to participate in the study (consent was obtained from the students,and proxy consent was obtained from guardians).

Exclusion Criteria There were no exclusion criteria for participation in this study.

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 360 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change in Depression Literacy measured by Depression Literacy Questionnaire (D-Lit) | is measured at baseline, directly after the intervention and three months follow-up.
  is measured by Depression Literacy Questionnaire (D-Lit)

SECONDARY OUTCOMES:
Change in Depression Stigma measured by Depression Stigma Scale (DSS) | is measured at baseline, directly after the intervention and three months follow-up.
  is measured by Depression Stigma Scale (DSS)
Change in Depression Self-Stigma measured by Self Stigma of Depression Scale (SSDS) | is measured at baseline, directly after the intervention and three months follow-up.
  is measured by Self Stigma of Depression Scale (SSDS)

CONTACTS AND LOCATIONS:
Locations (1):
- Jazan Education Sector, Jizan, Saudi Arabia